CLINICAL TRIAL: NCT06365372
Title: Circulating MrgD Change in Patients With Pulmonary Hypertension
Brief Title: Circulating MrgD in Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Professor, Qilu Hospital of Shandong University
Other Study IDs: MrgD and PAH
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAH
  Interventions: Diagnostic Test: Western blot
- Non-PAH
  Interventions: Diagnostic Test: Western blot

INTERVENTIONS:
Diagnostic Test: Western blot — Samples were measured by Western blot using a solution for the separation of lymphocytes from peripheral blood.

SUMMARY:
The aim of the study is to observe the change of the circulating MrgD level in patients with pulmonary hypertension compared with subjects without pulmonary hypertension.

ELIGIBILITY:
Inclusion criteria for patients with pulmonary hypertension：

1. Male or female aged ≥18 years
2. Right heart catheterisation to check the mean pulmonary artery pressure (mPAP) ≥25mmHg
3. The patient is willing and able to provide written informed consent.

Exclusion criteria for patients with pulmonary hypertension：

1. Age less than 18 years old
2. Mean pulmonary artery pressure (mPAP) <25mmHg
3. Unable to provide informed written consent for participation in the study
4. Renal insufficiency
5. Liver insufficiency
6. Malignant tumor
7. Active infection
8. Pregnancy

Inclusion criteria for control subjects：

1. Male or female aged ≥18 years
2. No evidence of pulmonary hypertension on echocardiography or mean pulmonary artery pressure (mPAP) < 25 mmHg on right heart catheterization, and no evidence of clinically relevant heart disease
3. No evidence of clinically relevant pulmonary disease

Exclusion criteria for control subjects：

1. Age less than 18 years old
2. Mean pulmonary artery pressure (mPAP) ≥25mmHg
3. Unable to provide informed written consent for participation in the study
4. Symptoms of heart failure or clinically relevant lung disease
5. Renal insufficiency
6. Liver insufficiency
7. Malignant tumor
8. Active infection
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension and control subjects
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Circulating MrgD level | From 2022 to 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided